CLINICAL TRIAL: NCT00116948
Title: A Comparison of Two Total Hip Replacements: Hip Resurfacing System Versus Mallory-Head/Exeter
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Biomet Merck Aps,Horsens, Denmark (Unknown); Gigtforeningen (Other); Sahva A/S, Borgervænget 5-7, København Ø, Denmark (Unknown); Danske Fysioterapeuter (Other); Regionshospitalet Silkeborg (Other); Finnish Institute of Occupational Health (Other); Regionshospitalet Hammel Neurocenter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20030289
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2014-12

CONDITIONS: Osteoarthrosis
Keywords: Osteoarthrosis; RSA; DEXA; Hip arthroplasty; Metal ion; Inflammatory response; Gait analysis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ReCap, Hip resurfacing system, Biomet — ReCap total hip arthroplasty inserted according to manufactures manual.

SUMMARY:
The purpose of this study is to compare two total hip replacement systems: Hip Resurfacing System (ReCap) versus Mallory-Head/Exeter.

DETAILED DESCRIPTION:
In Denmark approximately 7000 primary hip replacements are implanted yearly, and the incidence is rising with the increasingly aging population. For older patients, the incidence of later revisions of hip implantation is low. Unfortunately, this is not true for younger patients. Approximately 20% of patients under 55 years of age at the time of surgery must have the hip implant renewed within 10 years.

This is primarily because of the wear generated by polyethylene debris. The polyethylene is associated with osteolysis in the proximity of the prosthesis leading to failure of the prosthesis.

This unsatisfactory result has led to the development of an alternative hip prosthesis especially to benefit younger and physically active people. The new prosthesis should produce less inflammatory debris and less osteolysis induced failure.

To avoid the polyethylene particles, a new type of prosthesis has been made articulating metal on metal. The Hip Resurfacing System consists of an alloy of chrome - cobalt - molybdenum. Another point of interest for this prosthesis is also the size of the articulating surfaces which are bigger than usual. This will theoretically participate in the generation of metal ions.

Study objectives:

* This randomised prospective study will investigate the emission of Co-, Cr- and Mb-ions from Hip Resurfacing System and Mallory-Head/Exeter implants, respectively. The emission is measured as the ion concentration in the urine and is correlated to the inflammatory response in fasting plasma before and after the operation.
* To assess the walking pattern postoperatively using a 3D gait analysis, Vicon Polygon.
* To assess the postoperative recovery using the Harris hip score and visual analogue scale.
* The migration of acetabular components will be evaluated by RSA, performing radiostereometric analyses at the Orthopaedic Center, Aarhus University Hospital. The follow-up RSA will be scheduled for week 1, as well as 3 months, 12 months, 24 months, and 5 years after surgery. Bone mineral density around the implanted femoral component will be examined by DEXA scan at week 1, as well as 1 year and 2 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with primary hip osteoarthrosis (OA).
* Informed patient consent in writing.
* Sufficient bone density to allow uncemented implantation of an acetabular component.

Exclusion Criteria:

* Presence of other metal implants.
* Working exposure of chrome, cobalt or molybdenum.
* Ingestion of multivitamin or medication containing chrome, cobalt or molybdenum.
* Kidney disease
* Hip joint dysplasia
* Patients with neuromuscular or vascular disease in the affected leg.
* Patients who regularly take non-steroid anti-inflammatory drugs (NSAID) and cannot interrupt intake for the postoperative phase of the study.
* Patients with fracture sequelae.
* Female patients of childbearing capacity.
* Sequelae to previous hip joint disorder in childhood

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-01; Primary Completion 2011-09 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Metal ion release evaluated in urine | three years
Gait pattern evaluated with 3D gait analysis, Vicon Polygon | two years
Bone mineral density (BMD) in surrounding bone of the prosthesis | three years
Prostheses migration evaluated by radiostereometric analysis (RSA) | three years
Proinflammatory- and bone degradation measures in blood samples | three years

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Søballe, MD., Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Jylland, Denmark